CLINICAL TRIAL: NCT02311114
Title: Program Evaluation of Telehomecare for Patients With Heart Failure or Chronic Obstructive Pulmonary Disease: TeLeCare (TLC) Study
Brief Title: Program Evaluation of Telehomecare: TeLeCare Study
Acronym: TLC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Murray Krahn, MD MSc, University of Toronto
Other Study IDs: 30158
Record Dates: First submitted 2014-06-27; First posted 2014-12-08 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Program Evaluation; Telehomecare; Chronic Obstructive Pulmonary Disease; Heart Failure; LHINs; Local Health Integrative Network; OTN; Ontario Telemedicine Network
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Telehomecare patients: Observational fieldwork, in depth interviews and surveys up to 4 times will be conducted.
  Interventions: Other: In Depth interview; Other: Observational fieldwork; Other: Survey
- Health care providers: In-Depth interviews, observational fieldwork and one time survey will be conducted.
  Interventions: Other: In Depth interview; Other: Observational fieldwork; Other: Survey
- Telehomecare administrators: In depth interviews will be conducted
  Interventions: Other: In Depth interview; Other: Observational fieldwork
- Telehomecare technicians: In-depth interviews, observational fieldwork will be conducted.
  Interventions: Other: In Depth interview; Other: Observational fieldwork

INTERVENTIONS:
Other: In Depth interview — In Depth interview will be conducted for 30-60 min using semi-structured questionnaire to assess participants experience with telehomecare program.
Other: Observational fieldwork — Observational fieldwork will conducted to observe everyday routine activities related to telehomecare. May last up to 1h per observation.
Other: Survey — Surveys with participants will be conducted using validated survey tools.
  Groups: Health care providers; Telehomecare patients

SUMMARY:
This study will evaluate the Telehomecare (THC) Program offered to patients with heart failure or chronic obstructive pulmonary disease across the Central West, Toronto Central and North East Local Health Integration Networks in Ontario. It will explore the opinions and experiences of patients, providers, technicians and administrators involved with THC Program in order to provide stakeholders with information about the processes and organizational factors impacting the program's adoption, the experiences of its participants, impact on patient outcomes, costs to the health-care system and who is benefiting the most from participating. These factors will be determined using semi-structured interviews, surveys, and observation of practices of everyone involved with THC. The study will also evaluate patient data to determine changes in patients' utilization of healthcare services.

DETAILED DESCRIPTION:
The program evaluation will consist of three components that will employ two research methods, qualitative and quantitative.

Comparative Practice Study (Qualitative) This study will explore how factors related to the technology, patients, providers and organizational structures and processes influence the adoption and implementation of THC across selected sites (including micro-, meso- and macro-systems) in Ontario. Ethnographic study, in-depth semi-structured interviews and documentation collection and review will be employed to explore, among other factors, the behaviours, communication patterns, workflows and tasks of health care providers and their interaction with patients. Interviewees will be selected using purposive sampling.

Descriptive Study (Quantitative) The patterns of THC use will be evaluated by conducting a descriptive study based on the data routinely collected by the Ontario Telemedicine Newtrok that tracks all encounters (i.e. telephone calls, remote patient monitoring data transmission, face to face visits) between patients and THC providers. A randomly selected subset of THC participants/caregivers will also complete validated structured questionnaires at up to four time points during program, baseline, one, two, and three months after enrollment. These are the Quality of Life Profile Measure (SF12), Quality of Life Preference Measure (EQ5D), Telemedicine Perception Questionnaire (TMPQ), Stanford self-efficacy scale and Client Satisfaction Questionnaire (CSQ-8). The providers of THC will also be asked to complete questionnaires; physicians will be asked to complete Penn State Physician Telehomecare Survey, whereas the nurses will be asked to complete a Nurse Satisfaction Survey.

ICES Linkage Study (Quantitative) Primary collected research data will be linked to the Institute for Clinical Evaluative Sciences (ICES) administrative databases. Outcomes (i.e. hospitalizations, primary care visits) of patients receiving or have received Telehomecare, will be assessed for a period of 6 months prior to enrolment, during the program and for up to 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

Patient

* The patient has a documented diagnosis of HF or COPD (with or without co-morbid conditions)
* The patient is a 'heavy user' of the health care system, characterized by any of the following:
* A minimum of one hospitalization for a respiratory or cardiac complaint in the past six months
* A minimum of two emergency department/urgent care center visits for a respiratory or cardiac complaint in the past six months
* Is receiving nursing services via CCAC
* Frequent visits to primary care provider in the past year
* The patient or informal caregiver (if applicable) is an adult (over 18 yrs) able and willing to provide informed consent.
* The patient or informal caregiver (if applicable) is fluent in English
* The patient or informal caregiver is able and willing to operate the THC equipment
* The patient lives in a residential (private home or retirement home) setting with an active landline
* The patient or informal caregiver have agreed to be contacted for evaluation of this program when consenting to participate in the Telehomecare program.

Health Care Provider

* Any health care provider who referred a patient to the telehomecare program
* Primary care providers of patients who are enrolled in the study
* Telehomecare nurses/physicians involved in the provision of care to patients enrolled in the telehomecare program
* For interviews and surveys telehomecare nurses/physicians must have 3 months experience with telehomecare

Technician, Administrators and/or Decision Makers

* Technicians involved in the set-up of telehomecare equipment at patients' homes.
* Administrators and/or Decision Makers of the THC program as a larger network of care such as Healthcare Program Managers, key members of the LHIN, OTN etc.

Exclusion Criteria:

Patient

* Less than 18 years of age
* Individuals without an established diagnosis of COPD or chronic HF
* Unable or unwilling to provide verbal informed consent
* Demonstrated non-adherence to the THC program
* The THC Clinician works with each patient on a case-by-case review to assess willingness to partner in their own care, and if the number of missed consultation appointments and reasons for demonstrate overall non-adherence with the program.
* Inability or unwillingness to use THC equipment
* Do not have a regular caregiver to assist in the use of the equipment

Health Care Provider, Technician, Administrators and/or Decision Makers

- Unable or unwilling to provide verbal informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care providers, technicians, administrators/decision makers and patients enrolled in the Telehomecare Program.
Sampling Method: Non-Probability Sample
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Organizational Factors (Semi-structured interviews and general observation) | The data collection period will be approximately 3 months
  Those factors will be identified via qualitative research methods, hence no measurable units are applicable for them.
  Semi-structured interviews and general observation of all types of participants will be done at different times/stages of program.

SECONDARY OUTCOMES:
Overall patterns of use (length of stay, drop out rates, nurse workload, etc.) | Retrospectively using Ontario Telemedicine Network database, for all participants who were enrolled in the Telehomecare program. The data collection period will be approximately 3 months
  Participants' demographics, average length of stay within the program, drop out rates, nurses workload (number of patients per nurses), number of alerts per patients and per nurse.
Telemedicine perception (Telemedicine perception questionnaire (TMPQ)) | Prospectively at baseline, and at month 1, 2, 3 follow-up
  Measured via Telemedicine perception questionnaire (TMPQ)
Health services utilization (hospitalization, LOS, ED visits, etc.) | Retrospectively, six months before, during and after the Telehomecare program. Will be collected for the patients who completed the Telehomecare by the 28 Feb 2014.
  Number of hospitalizations, length of stay, ED visits, primary care visits, cost related to health services utilization. Will be done through linkage with ICES database
Quality of life | Prospectively at baseline, and at month 1, 2, 3 follow-up
  Measured via EQ-5D and SF-12 questionnaires
Client satisfaction (satisfaction questionnaire (CSQ-8) | Prospectively at baseline, and at month 1, 2, 3 follow-up
  Measured via client satisfaction questionnaire (CSQ-8)
Chronic disease management (Stanford Chronic Disease Self-Management 33-item scale) | Prospectively at baseline, and at month 1, 2, 3 follow-up
  Measured via Stanford Chronic Disease Self-Management 33-item scale

CONTACTS AND LOCATIONS:
Overall Officials: Murray Krahn, MD,MSc, Principal Investigator — THETA Collaborative; Valeria Rac, MD, PhD, Principal Investigator — THETA Collaborative
Locations (1):
- University of Toronto, Toronto, Canada